CLINICAL TRIAL: NCT05271513
Title: The Use of Non-invasive Trans-spinal Magnetic Stimulation to Enhance the Efficacy of Trans-cranial Magnetic Stimulation in Advanced PD With Axial Motor Symptoms: Double Blinded Randomized Clinical Trial
Brief Title: Efficacy of Repetitive Trans-spinal Magnetic Stimulation on Axial Motor Symptoms in PD
Acronym: rTSMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rTSMS in Parkinson's disease
Record Dates: First submitted 2021-12-26; First posted 2022-03-09 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Adverse Effect of Drug Therapy Levodopa
Keywords: rTMS; Parkinson's disease; therapeutic role; spinal magnetic stimulation; gait disturbance, frozen gait; UPDRS, Quality of life, Visual analogue scale
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: masking enclosed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real transcranial magnetic stimulation plus real transcutaneous magnetic stimulation of spinalcord (Active Comparator): the patient will receive real rTMS 2000 pulses for each hand area 20Hz 80% of Motor threshold of the hand, 10 trains, each train 10 seconds over the hand area plus 1000 pulses 10 Hz 80% of the motor threshold of the leg 10 trains, and each train 10 seconds over the mid-cervical vertebrae for consecuative 10 days (5 days/week)
  Interventions: Device: non invasive repetitive magnetic stimulation (real Transcranial + real trans-spinal )
- real transcranial magnetic stimulation with sham transcutaneous magnetic stimulation of spinalcord (Active Comparator): the patient will receive real rTMS 2000 pulses for each hand area 20Hz 80% of Motor threshold of the hand, 10 trains, each train 10 seconds plus sham stimulation 1000 pulses 10 Hz 80% of the motor threshold of the leg 10 trains, and each train 10 seconds over the mid-dorsal vertebrae for 10 consecutive days (5 sessions/week)
  Interventions: Device: non invasive repetitive magnetic stimulation (real Transcranial + sham trans-spinal )sham trans-spinal magnetic stimulation

INTERVENTIONS:
Device: non invasive repetitive magnetic stimulation (real Transcranial + real trans-spinal ) — repetitive transcranial magnetic stimulation and trans-spinal magnetic stimulation
  Arms: real transcranial magnetic stimulation plus real transcutaneous magnetic stimulation of spinalcord
Device: non invasive repetitive magnetic stimulation (real Transcranial + sham trans-spinal )sham trans-spinal magnetic stimulation — sham trans-spinal magnetic stimulation
  Arms: real transcranial magnetic stimulation with sham transcutaneous magnetic stimulation of spinalcord

SUMMARY:
The purpose of this randomized trial was to evaluate the efficacy of repeated sessions of trans-spinal magnetic stimulation on gait abnormality, and posture abnormalities in patients with idiopathic Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease is the second most common age-related neurodegenerative disease after Alzheimer's disease[1], patients with advanced Parkinson's disease (PD) often present with axial symptoms, including abnormal posture, postural instability, and gait disorder [2]. These axial symptoms are the main factors that reduce the activities of daily living (ADL) and quality of life (QOL) of PD patients. Gait disorders are among the most prevalent problems in the advanced phase of Parkinson's disease (PD) and are relatively resistant to dopaminergic treatment. Freezing of gait (FoG) affects 7% of patients in early PD and reaches 60% in advanced stages [3]. Patients with PD also suffer from pain significantly more frequently than normal subjects. Low back pain and leg pain are the most commonly experienced pain symptoms in PD patients. One of the reasons is considered to be the decreased threshold of pain due to abnormality of the dopaminergic system in the basal ganglia of PD patients [3.4]. Administration of anti-parkinsonian medication or Deep brain stimulation results in increased pain thresholds. Treatment by medication or DBS is often ineffective for low back pain caused by postural deformity and is also ineffective for radicular or peripheral neuropathic. Because pain is an important factor that reduces the ADL and QOL of patients, the establishment of new and effective therapy is essential [5.6]. A positive effect of epidural spinal cord stimulation (SCS) on locomotive activity has been reported in animal models and small cohorts of PD patients and seems to be promising.[7] Transcutaneous SCS is an emerging method that activates similar target neural structures noninvasively and has recently been explored for the treatment of spasticity after spinal cord injury.[8] Here, the investigators will assess the safety and efficacy of transcutaneous magnetic SCS on freezing of gait (FoG) and other motor symptoms in a cohort of PD patients.

The investigators will be going to carry out a double-blinded randomized, case-controlled study on 42 patients who will be randomly chosen and categorize them into 2 groups, 21 patients each. The 1st group will receive real transcranial magnetic stimulation applied over each hand area High frequency 20 HZ, 80% of the motor threshold of hand, 10 sec for each train, 20 train with a total of 2000 pulses for each side plus transcutaneous spinal cord stimulation (over mid-dorsal vertebrae (thoracic 6) high frequency 10 HZ, 80% of the motor threshold of leg area10 sec for each train, 10 trains with total 1000 pulses for 10 consecutive days. The second group will receive the same protocol but the spinal stimulation will be sham stimulation as the coil lie perpendicular to the vertebral axis. Then the investigators will be going to compare the results of two groups at the end of sessions, one and two months after the last session to find out the efficacy of repetitive transcutaneous magnetic stimulation of the spinal cord on gait abnormalities and posture abnormalities, relief of pain, UPDRS, and as well as the quality of life in patients with idiopathic Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

1. Men or women of at least 40-80 years of age.
2. Are reliable and willing to make themselves available for the duration of the study and are willing to follow up.
3. Medically stable outpatients with a confirmed diagnosis of idiopathic PD according to United Kingdom Brain Bank Criteria
4. Clear written informed consent from each participant in the trial.
5. Patients after at least 6 h free of parkinsonian drugs (off-state).

Exclusion Criteria:

1. Pregnants, breastfeeding, or willing to be pregnant during the study.
2. Presence of a clinically significant medical or psychiatric condition that may increase the risk associated with the study
3. Participation in any other type of medical research that may interfere with the interpretation of the study.
4. Patients with severe motor disability (bed-ridden ) that may interfere with the study procedure.
5. History of surgical or invasive intervention for Parkinson's disease.
6. Patients with a history of seizures or epilepsy including history in a first-degree relative or patients on treatment that reduce the seizure threshold.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Score on Freezing of gait Questionnaire | 2 months after the end of sessions
  Score on Freezing of gait Questionnaire
Time taken for Primed up-and-go | 2 months after the end of sessions
  Time taken for Primed up-and-go
Time taken for 10m walk | 2 months after the end of sessions
  Time taken for 10m walk

SECONDARY OUTCOMES:
Score on MDS-UPDRS | 2 months after the end of sessions
  Score on MDS-UPDRS
Score on PDQ-39 | 2 months after the end of sessions
  Score on PDQ-39

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Fuentes R, Petersson P, Nicolelis MA. Restoration of locomotive function in Parkinson's disease by spinal cord stimulation: mechanistic approach. Eur J Neurosci. 2010 Oct;32(7):1100-8. doi: 10.1111/j.1460-9568.2010.07417.x. PMID 21039949
- [Background] Doherty KM, van de Warrenburg BP, Peralta MC, Silveira-Moriyama L, Azulay JP, Gershanik OS, Bloem BR. Postural deformities in Parkinson's disease. Lancet Neurol. 2011 Jun;10(6):538-49. doi: 10.1016/S1474-4422(11)70067-9. Epub 2011 Apr 22. PMID 21514890
- [Background] Fuentes R, Petersson P, Siesser WB, Caron MG, Nicolelis MA. Spinal cord stimulation restores locomotion in animal models of Parkinson's disease. Science. 2009 Mar 20;323(5921):1578-82. doi: 10.1126/science.1164901. PMID 19299613
- [Background] Moorehead MK, Ardelt-Gattinger E, Lechner H, Oria HE. The validation of the Moorehead-Ardelt Quality of Life Questionnaire II. Obes Surg. 2003 Oct;13(5):684-92. doi: 10.1381/096089203322509237. PMID 14627461
- [Result] Poewe W, Seppi K, Tanner CM, Halliday GM, Brundin P, Volkmann J, Schrag AE, Lang AE. Parkinson disease. Nat Rev Dis Primers. 2017 Mar 23;3:17013. doi: 10.1038/nrdp.2017.13. PMID 28332488
- [Result] Agari T, Date I. Spinal cord stimulation for the treatment of abnormal posture and gait disorder in patients with Parkinson's disease. Neurol Med Chir (Tokyo). 2012;52(7):470-4. doi: 10.2176/nmc.52.470. PMID 22850494
- [Result] Defazio G, Berardelli A, Fabbrini G, Martino D, Fincati E, Fiaschi A, Moretto G, Abbruzzese G, Marchese R, Bonuccelli U, Del Dotto P, Barone P, De Vivo E, Albanese A, Antonini A, Canesi M, Lopiano L, Zibetti M, Nappi G, Martignoni E, Lamberti P, Tinazzi M. Pain as a nonmotor symptom of Parkinson disease: evidence from a case-control study. Arch Neurol. 2008 Sep;65(9):1191-4. doi: 10.1001/archneurol.2008.2. PMID 18779422
- [Result] Djaldetti R, Shifrin A, Rogowski Z, Sprecher E, Melamed E, Yarnitsky D. Quantitative measurement of pain sensation in patients with Parkinson disease. Neurology. 2004 Jun 22;62(12):2171-5. doi: 10.1212/01.wnl.0000130455.38550.9d. PMID 15210877
- [Result] Brefel-Courbon C, Payoux P, Thalamas C, Ory F, Quelven I, Chollet F, Montastruc JL, Rascol O. Effect of levodopa on pain threshold in Parkinson's disease: a clinical and positron emission tomography study. Mov Disord. 2005 Dec;20(12):1557-63. doi: 10.1002/mds.20629. PMID 16078219
- [Result] Gerdelat-Mas A, Simonetta-Moreau M, Thalamas C, Ory-Magne F, Slaoui T, Rascol O, Brefel-Courbon C. Levodopa raises objective pain threshold in Parkinson's disease: a RIII reflex study. J Neurol Neurosurg Psychiatry. 2007 Oct;78(10):1140-2. doi: 10.1136/jnnp.2007.120212. Epub 2007 May 15. PMID 17504881
- [Result] Yadav AP, Nicolelis MAL. Electrical stimulation of the dorsal columns of the spinal cord for Parkinson's disease. Mov Disord. 2017 Jun;32(6):820-832. doi: 10.1002/mds.27033. Epub 2017 May 12. PMID 28497877
- [Result] Hofstoetter US, Freundl B, Danner SM, Krenn MJ, Mayr W, Binder H, Minassian K. Transcutaneous Spinal Cord Stimulation Induces Temporary Attenuation of Spasticity in Individuals with Spinal Cord Injury. J Neurotrauma. 2020 Feb 1;37(3):481-493. doi: 10.1089/neu.2019.6588. Epub 2019 Aug 9. PMID 31333064
- [Result] Postuma RB, Poewe W, Litvan I, Lewis S, Lang AE, Halliday G, Goetz CG, Chan P, Slow E, Seppi K, Schaffer E, Rios-Romenets S, Mi T, Maetzler C, Li Y, Heim B, Bledsoe IO, Berg D. Validation of the MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2018 Oct;33(10):1601-1608. doi: 10.1002/mds.27362. Epub 2018 Aug 25. PMID 30145797
- [Derived] Khedr EM, Haridy NA, Korayem MA, Tawfik AM, Hamed AA. In PD, Non-Invasive Trans-Spinal Magnetic Stimulation Enhances the Effect of Transcranial Magnetic Stimulation on Axial Motor Symptoms: A Double-Blind Randomized Clinical Trial. Neurorehabil Neural Repair. 2025 Feb;39(2):126-137. doi: 10.1177/15459683241300547. Epub 2024 Dec 11. PMID 39659276